CLINICAL TRIAL: NCT06107218
Title: Performance Of Occlusal Resin Composite Restorations Following Cavity Finishing Using Bioactive Glass Air Abrasion Versus Diamond Stone: A Randomized Controlled Trial
Brief Title: Performance Of Class I Composite Restorations After Cavity Finishing By Air Abrasion Versus Diamond Stone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Essam Mahmoud, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Air Abrasion in Finishing
Record Dates: First submitted 2023-10-10; First posted 2023-10-30 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Abrasion, Dental; Class I Dental Caries
MeSH Terms: conditions — Tooth Abrasion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diamond Stone group (Comparator) (Active Comparator): Class I cavities will be finished using 20-30 μm grit extra fine (EF) yellow coded diamond stone with maximum rotational speed 300,000 min -1.
  Interventions: Other: Diamond Stone.
- Bioactive Glass Air Abrasion group (Intervention) (Active Comparator): Class I cavities will be finished by AquaCare Air Abrasion Device using bioactive glass air-abrasion particles (a mix of 30-60-90 μm particles). The nozzle of the air abrasion device will be 0.6 in diameter and angulated at 90° to the occlusal surface with a distance away from the tooth about 2-3 mm. The device will be used in a dynamic motion with 60 psi (4 Bar) adjusted pressure for 3 seconds.
  Interventions: Other: Bioactive Glass Air Abrasion Particles.

INTERVENTIONS:
Other: Bioactive Glass Air Abrasion Particles. — Finishing of cavity walls by AquaCare Air Abrasion Device using Bioactive Glass Air Abrasion Particles.
  Arms: Bioactive Glass Air Abrasion group (Intervention)
Other: Diamond Stone. — Finishing of cavity walls using Diamond Stone.
  Arms: Diamond Stone group (Comparator)

SUMMARY:
The aim of the study is to reveal the performance of the resin composite restorations after finishing the cavity walls and margins using bioactive glass air abrasion particles in comparison to the routine finishing with the finishing diamond stone according to the FDI criteria for post operative sensitivity, marginal adaptation, marginal discoloration, secondary caries, and retention.

DETAILED DESCRIPTION:
Intraoral air abrasion is the process of altering the surface of the tooth structure through the use of abrasive particles propelled by compressed air or other gasses. The use of intraoral air abrasion has become practical with devices that simultaneously output abrasive particles and water to control the spread of the particles. There are different types of abrasive particles maybe used depending on the clinical application for which the intraoral air abrasion is being performed. Intraoral air abrasion may also be used as a tool for dental prophylaxis, often called air polishing.

Different particles could be incorporated into air abrasion devices according to the intended use of them, such as aluminum oxide (alumina), Calcium Sodium Phosphosilicate (Biactive Glass) and Sodium bicarbonate. To obtain maximum cutting efficiency, the particle should be hard enough to indent the substrate it abrades, and irregular in shape with a sharp cutting edge. Round and smooth particles possess poor abrasive properties, so it may be used for polishing needs "air- polishing". Increased air pressure provided an increased number and velocity of the particles. Abrading power must be proportional to kinetic energy of the particles, which is the function of mass and velocity of the particle. The cutting efficiency of air abrasion depends on several criteria, such as: size, shape, hardness, density of the particles and air pressure.

Aluminum oxide (alumina) are the most abrasive type of particles used. They are irregular in shape with different particle sizes. Intraoral sandblasting with alumina particles (Al2O3) was first described in 1945 by Black. Initially, it was reported that the bond strength to the tooth surface improved, also confirmed by recent investigations, and some authors adopted its use in clinical procedures even after preparing the cavity with rotating instrument. A bioactive glass abrasive, is also commercially available but indicated for the purpose of tooth polishing. Some work has also showed potential for it to have selective cutting properties. However, its cutting time can take 2-3 times longer than alumina, making it clinically indicated for cavity finishing and not cutting.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene (plaque index score 0 or 1).
* Absence of abnormal occlusion habits (e.g. bruxism, nail biting, tooth clenching and mouth breathing).
* Patients approving to participate in the study.

Exclusion Criteria:

* Patients with known allergic or adverse reaction to the tested materials.
* Systematic disease that may affect participation.
* Xerostomic patients.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Post-operative sensitivity. | 24 hours Baseline, 6 and 12 months.
  The restorations will be assessed and evaluated by Visual Analogue Scale using Federation Dentaire Internationale (FDI) criteria. Visual Analogue Scale will be used by scores ranging from 0 to 10, where 0 indicates no pain and 10 indicates maximum pain.

SECONDARY OUTCOMES:
Marginal Discoloration. | 24 hours Baseline, 6, 12 and 18 months.
  The restorations will be assessed by visual examination and short air drying. Assessment will be done using FDI criteria and recorded as scores from 1 to 5, where scores from 1 to 5 will indicate clinically excellent/very good, clinically good, clinically satisfactory, clinically unsatisfactory and clinically poor respectively.
Marginal Adaptation. | 24 hours Baseline, 6, 12 and 18 months.
  The Method of restorations assessment will be Tactile using different sized explorers. Assessment will be done using FDI criteria and recorded as scores from 1 to 5, where scores from 1 to 5 will indicate clinically excellent/very good, clinically good, clinically satisfactory, clinically unsatisfactory and clinically poor respectively.
Occurrence of Caries. | 24 hours Baseline, 6, 12 and 18 months.
  The Method of restorations assessment will be Tactile using different sized explorers. Assessment will be done using FDI criteria and recorded as scores from 1 to 5, where scores from 1 to 5 will indicate clinically excellent/very good, clinically good, clinically satisfactory, clinically unsatisfactory and clinically poor respectively.
Loss of Retention. | 24 hours Baseline, 6, 12 and 18 months.
  The restorations will be assessed by visual examination and short air drying. Assessment will be done using FDI criteria and recorded as scores from 1 to 5, where scores from 1 to 5 will indicate clinically excellent/very good, clinically good, clinically satisfactory, clinically unsatisfactory and clinically poor respectively.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang CT, Kim J, Arce C, Lawson NC. Intraoral Air Abrasion: A Review of Devices, Materials, Evidence, and Clinical Applications in Restorative Dentistry. Compend Contin Educ Dent. 2019 Sep;40(8):508-513; quiz 514. PMID 31478697
- [Background] Paolinelis G, Banerjee A, Watson TF. An in vitro investigation of the effect and retention of bioactive glass air-abrasive on sound and carious dentine. J Dent. 2008 Mar;36(3):214-8. doi: 10.1016/j.jdent.2007.12.004. Epub 2008 Jan 30. PMID 18237840
- [Background] Banerjee A, Pabari H, Paolinelis G, Thompson ID, Watson TF. An in vitro evaluation of selective demineralised enamel removal using bio-active glass air abrasion. Clin Oral Investig. 2011 Dec;15(6):895-900. doi: 10.1007/s00784-010-0470-2. Epub 2010 Oct 13. PMID 20941634
- [Background] Banerjee A, Thompson ID, Watson TF. Minimally invasive caries removal using bio-active glass air-abrasion. J Dent. 2011 Jan;39(1):2-7. doi: 10.1016/j.jdent.2010.09.004. Epub 2010 Oct 1. PMID 20888883
- [Background] Milly H, Austin RS, Thompson I, Banerjee A. In vitro effect of air-abrasion operating parameters on dynamic cutting characteristics of alumina and bio-active glass powders. Oper Dent. 2014 Jan-Feb;39(1):81-9. doi: 10.2341/12-466-L. Epub 2013 May 29. PMID 23718212
- [Background] Lynch CD, Opdam NJ, Hickel R, Brunton PA, Gurgan S, Kakaboura A, Shearer AC, Vanherle G, Wilson NH; Academy of Operative Dentistry European Section. Guidance on posterior resin composites: Academy of Operative Dentistry - European Section. J Dent. 2014 Apr;42(4):377-83. doi: 10.1016/j.jdent.2014.01.009. Epub 2014 Jan 22. PMID 24462699
- [Background] da Rosa Rodolpho PA, Cenci MS, Donassollo TA, Loguercio AD, Demarco FF. A clinical evaluation of posterior composite restorations: 17-year findings. J Dent. 2006 Aug;34(7):427-35. doi: 10.1016/j.jdent.2005.09.006. Epub 2005 Nov 28. PMID 16314023
- [Background] Hofsteenge JW, Scholtanus JD, Ozcan M, Nolte IM, Cune MS, Gresnigt MMM. Clinical longevity of extensive direct resin composite restorations after amalgam replacement with a mean follow-up of 15 years. J Dent. 2023 Mar;130:104409. doi: 10.1016/j.jdent.2023.104409. Epub 2023 Jan 6. PMID 36623686
- [Background] Hardan L, Sidawi L, Akhundov M, Bourgi R, Ghaleb M, Dabbagh S, Sokolowski K, Cuevas-Suarez CE, Lukomska-Szymanska M. One-Year Clinical Performance of the Fast-Modelling Bulk Technique and Composite-Up Layering Technique in Class I Cavities. Polymers (Basel). 2021 Jun 4;13(11):1873. doi: 10.3390/polym13111873. PMID 34200021
- [Background] Van Meerbeek B, De Munck J, Mattar D, Van Landuyt K, Lambrechts P. Microtensile bond strengths of an etch&rinse and self-etch adhesive to enamel and dentin as a function of surface treatment. Oper Dent. 2003 Sep-Oct;28(5):647-60. PMID 14531614
- [Background] Graumann SJ, Sensat ML, Stoltenberg JL. Air polishing: a review of current literature. J Dent Hyg. 2013 Aug;87(4):173-80. PMID 23986410
- [Background] Bendinskaite R, Peciuliene V, Brukiene V. A five years clinical evaluation of sealed occlusal surfaces of molars. Stomatologija. 2010;12(3):87-92. PMID 21063138
- [Background] Cvar JF, Ryge G. Reprint of criteria for the clinical evaluation of dental restorative materials. 1971. Clin Oral Investig. 2005 Dec;9(4):215-32. doi: 10.1007/s00784-005-0018-z. No abstract available. PMID 16315023
- [Background] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Science Committee Project 2/98--FDI World Dental Federation study design (Part I) and criteria for evaluation (Part II) of direct and indirect restorations including onlays and partial crowns. J Adhes Dent. 2007;9 Suppl 1:121-47. PMID 18341239
- [Background] Marquillier T, Domejean S, Le Clerc J, Chemla F, Gritsch K, Maurin JC, Millet P, Perard M, Grosgogeat B, Dursun E. The use of FDI criteria in clinical trials on direct dental restorations: A scoping review. J Dent. 2018 Jan;68:1-9. doi: 10.1016/j.jdent.2017.10.007. Epub 2017 Oct 18. PMID 29055692
- [Background] Hickel R, Mesinger S, Opdam N, Loomans B, Frankenberger R, Cadenaro M, Burgess J, Peschke A, Heintze SD, Kuhnisch J. Revised FDI criteria for evaluating direct and indirect dental restorations-recommendations for its clinical use, interpretation, and reporting. Clin Oral Investig. 2023 Jun;27(6):2573-2592. doi: 10.1007/s00784-022-04814-1. Epub 2022 Dec 12. PMID 36504246
- [Background] Martinez-Insua A, Da Silva Dominguez L, Rivera FG, Santana-Penin UA. Differences in bonding to acid-etched or Er:YAG-laser-treated enamel and dentin surfaces. J Prosthet Dent. 2000 Sep;84(3):280-8. doi: 10.1067/mpr.2000.108600. PMID 11005900
- [Background] Turkistani A, Almutairi M, Banakhar N, Rubehan R, Mugharbil S, Jamleh A, Nasir A, Bakhsh T. Optical Evaluation of Enamel Microleakage with One-Step Self-Etch Adhesives. Photomed Laser Surg. 2018 Nov;36(11):589-594. doi: 10.1089/pho.2018.4441. Epub 2018 May 29. PMID 29813001
- [Background] Torres CRG, Mailart MC, Crastechini E, Feitosa FA, Esteves SRM, Di Nicolo R, Borges AB. A randomized clinical trial of class II composite restorations using direct and semidirect techniques. Clin Oral Investig. 2020 Feb;24(2):1053-1063. doi: 10.1007/s00784-019-02999-6. Epub 2019 Jul 9. PMID 31290018
- [Background] Nemt-Allah AA, Ibrahim SH, El-Zoghby AF. Marginal Integrity of Composite Restoration with and without Surface Pretreatment by Gold and Silver Nanoparticles vs Chlorhexidine: A Randomized Controlled Trial. J Contemp Dent Pract. 2021 Oct 1;22(10):1087-1097. PMID 35197374
- [Background] Paula EA, Tay LY, Kose C, Mena-Serrano A, Reis A, Perdigao J, Loguercio AD. Randomized clinical trial of four adhesion strategies in cervical lesions: 12-month results. Int J Esthet Dent. 2015 Spring;10(1):122-145. PMID 25625130
- [Background] Perdigao J, Kose C, Mena-Serrano AP, De Paula EA, Tay LY, Reis A, Loguercio AD. A new universal simplified adhesive: 18-month clinical evaluation. Oper Dent. 2014 Mar-Apr;39(2):113-27. doi: 10.2341/13-045-C. Epub 2013 Jun 26. PMID 23802645